CLINICAL TRIAL: NCT02906410
Title: Dynamic Presentation of Calorie Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Eric VanEpps, Postdoctoral Fellow, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Dynamic Presentation
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Not Condition-specific

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Control 1 (No Intervention): Participants in this group will see a menu labeled with prices, but will not observe calorie information. Used as a comparator for numeric labeling conditions.
- Numeric individual (Experimental): Features Item-Level Calorie information. Numeric calorie labels will be featured on individual items, along with prices.
  Interventions: Other: Item-Level Calorie information
- Numeric individual + aggregate (Experimental): Features Item-Level Calorie information and Meal-Level Calorie information. Numeric calorie labels will be featured on individual items, along with prices. Additionally, an aggregated numeric calorie count for the entire meal will be dynamically updated as items are added or removed from the meal.
  Interventions: Other: Item-Level Calorie information; Other: Meal-Level Calorie information
- Control 2 (No Intervention): Participants in this group will see a menu labeled with prices, but will not observe calorie information. Used as a comparator for light labeling conditions.
- Light individual (Experimental): Features Item-Level Calorie information. Traffic light calorie labels will be featured on individual items, along with prices.
  Interventions: Other: Item-Level Calorie information
- Light individual + aggregate (Experimental): Features Item-Level Calorie information and Meal-Level Calorie information. Traffic light calorie labels will be featured on individual items, along with prices. Additionally, an aggregated traffic light label for the entire meal will be dynamically updated as items are added or removed from the meal.
  Interventions: Other: Item-Level Calorie information; Other: Meal-Level Calorie information

INTERVENTIONS:
Other: Item-Level Calorie information — Information identifying the calorie content of individual items will be provided, as would be done on a restaurant menu board.
  Arms: Light individual; Light individual + aggregate; Numeric individual; Numeric individual + aggregate
Other: Meal-Level Calorie information — Information from the calorie content of individual items that have been selected by the participant will be dynamically aggregated and presented as a "Total Calories" label on the menu screen.
  Arms: Light individual + aggregate; Numeric individual + aggregate

SUMMARY:
Participants will be asked to select a hypothetical lunch from a menu that features entrees, sides, and drinks. Participants will be able to select a maximum of 1 item from each category. Following this meal selection, participants will complete a short survey about their demographics, their estimates of information about the meal and about recommended eating habits.

DETAILED DESCRIPTION:
The presence or absence of calorie labels on the hypothetical lunch menu will be randomly assigned to participants. Participants will first be randomly assigned to either the numeric label survey or the light label survey, and then within that survey, participants will be randomly assigned to either a control (no label), an item-level label, or an item-level and meal-level label condition.

Participants will select a hypothetical lunch from a menu that features entrees, sides, and drinks. Participants will be able to select a maximum of 1 item from each category. Following this meal selection, participants will complete a short survey about their demographics, their estimates of information about the meal and about recommended eating habits.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* US resident

Exclusion Criteria:

* Unable to complete survey on computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8544 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Calories ordered | 5 minutes after presentation of information
  Single survey presentation, measure of calories ordered collected as people select meal

SECONDARY OUTCOMES:
Light category ordered | 5 minutes after presentation of information
  Single survey presentation, measure of what aggregated light the calories ordered would have qualified for. Collected as people select meal
Calories per category | 5 minutes after presentation of information
  Single survey presentation, measure of calories per entree, calories per side, and calories per drink selected, collected as people select meal

OTHER OUTCOMES:
Sequence of items selected | 5 minutes after presentation of information
  Single survey presentation, measure of which items were added (and subtracted) from the meal. Both offers a count of number of items considered and a measure of calories "removed" from meal.

CONTACTS AND LOCATIONS:
Overall Officials: Eric VanEpps, PhD, Principal Investigator — Postdoctoral Fellow

IPD SHARING:
Plan to Share IPD: Undecided